CLINICAL TRIAL: NCT06370468
Title: To Elucidate the Epidemiological, Clinical, and Intrinsic Characteristics of Chronic Rhinitis
Brief Title: The Epidemiological and Intrinsic Characteristics of Chronic Rhinitis
Status: Recruiting | Type: Observational
Sponsor: Zheng Liu ENT (Other)
Collaborators: Peking Union Medical College (Other); Hainan People's Hospital (Other); Shandong Second Provincial General Hospital (Unknown); First Affiliated Hospital of Chongqing Medical University (Other); First Affiliated Hospital of Xinjiang Medical University (Other)
Responsible Party: Sponsor-Investigator, Zheng Liu ENT, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: 2024-CR-China
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Chronic Rhinitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum, blood cells, urine, nasal secretion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 18000 cases: The first part of the study will use a multi-stage cluster sampling survey, aiming to complete a questionnaire survey of 18,000 cases to assess the incidence and characteristics of chronic rhinitis. Each center will need to complete 3,000 face-to-face questionnaires to ensure reliable survey results.
  Interventions: Other: Epidemiological investigation
- 132000 cases: The second part will involve distributing 132,000 electronic questionnaires to community health service centers through convenient sampling. This method will allow us to obtain a large volume of questionnaire data more conveniently, thereby enhancing our investigation and analysis of chronic rhinitis. Each of the six centers will need to complete 22,000 online questionnaires.
  Interventions: Other: Epidemiological investigation

INTERVENTIONS:
Other: Epidemiological investigation — Epidemiological investigation

SUMMARY:
Chronic rhinitis affects 10-40% of China's population, or over 300 million people, and can lead to respiratory and psychological issues. Despite treatment progress, 30% of patients have poor outcomes, likely due to the disease's complexity and a lack of new treatment targets. The incidence is rising, but there's a lack of nationwide studies on its variations. This study addresses this through a multicentric survey to create a national database on chronic rhinitis, including epidemiological, clinical, and biological data. The goal is to understand chronic rhinitis's causes and risks, improve treatments, and develop preventive strategies. The study will survey 30,000 patients across China, using questionnaires and nasal exams, and preserve biological samples in a biobank for detailed analysis. This will lay the groundwork for understanding the disease's mechanisms, developing new diagnostics, and tailoring prevention and treatment approaches for different forms of chronic rhinitis.

DETAILED DESCRIPTION:
1. Epidemiological Investigation 1.1 Survey Group Selection: This study aims to conduct an epidemiological survey of chronic rhinitis across various regions of China, including the north, central, south, east, and west. The objective is to gather epidemiological, demographic, and clinical information from 30,000 patients with chronic rhinitis (5,000 cases per center) through questionnaires. Assuming a prevalence rate of chronic rhinitis at 20% of the population, approximately 150,000 questionnaires will be required. To ensure the project's efficiency and scientific rigor, it is divided into two parts. Initially, a multi-stage cluster random sampling survey will be conducted, encompassing 18,000 cases for a face-to-face questionnaire survey to accurately assess the incidence and characteristics of chronic rhinitis. Using a multi-stage cluster random sampling method, three administrative districts will be randomly selected from the central urban area of each city, one street from each district, and two residential areas from each street. Cluster sampling will be used to collect 500 questionnaire results from residents aged 18 to 70 in each residential area.

For the remaining 132,000 questionnaires, electronic questionnaires will be distributed to communities or community health service centers for online surveys using convenient sampling methods. Residents aged 18 to 70 will be encouraged to participate, and the data will be collected and analyzed.

1.2 Survey Indicators: Volunteers who respond positively to "whether they have chronic rhinitis" will be surveyed using a general information questionnaire and a chronic rhinitis-specific questionnaire.

The chronic rhinitis questionnaire primarily covers the following areas: living environment, symptoms experienced, medical history, and the pattern of disease manifestation (intermittent or persistent). It also inquires about the impact on daily life, including a severity assessment, potential predisposing factors, diagnostic methods employed (such as allergen testing), treatment approaches (including surgery, medication, and desensitization therapy), the level of disease control achieved, presence of any concurrent diseases, and the types of allergic conditions prevalent among family members.

Chronic rhinitis patients who successfully complete the face-to-face questionnaire and demonstrate good cooperation will be provided with a free nasal examination voucher and invited to the center for a specialist examination and the collection of corresponding biological specimens.

1.3 Specialist Examination and Biological Sample Collection:

* Serum sIgE or skin prick tests (SPT): SPT will be conducted to determine the presence of atopic constitution. The foundational allergen detection panel comprises the following allergens: dermatophagoides farinae, Dermatophagoides pteronyssinus, Artemisia vulgaris (mugwort), birch, Humulus lupulus (common hop), sycamore, cockroach, cat dander, dog dander, and Alternaria alternata (alternating Streptospora)." The SPT is typically conducted on the volar side of the forearm, and it necessitates the cessation of medications that could interfere with the results, such as antihistamines, for a period of 3 to 7 days prior to the test. During the procedure, both a histamine positive control and a saline negative control are utilized. The recommended concentration for the histamine positive control is 10 mg/ml. A wheal diameter exceeding 3 mm is considered indicative of a positive reaction in the SPT. The test results should be evaluated between 15 to 20 minutes after the application of the allergens. It is important to note that some individuals may exhibit delayed reactions, which require medical attention if they occur. Patients testing positive are diagnosed with Allergic Rhinitis (AR), while those testing negative proceed to the subsequent diagnostic step.
* Allergen nasal provocation (ANP): The ANP test is conducted to diagnose Local Allergic Rhinitis (LAR) by directly introducing allergens into the nasal cavity to induce nasal allergy symptoms. Here's a refined description of the procedure:

  1. Medication Suspension: Patients are instructed to cease the use of any medications that might interfere with the test outcomes, such as antihistamines and corticosteroid nasal sprays, typically for a period exceeding 48 hours prior to the test.
  2. Patient Evaluation: A comprehensive health assessment is performed to ensure that the patient does not exhibit severe nasal congestion or acute respiratory infections, as these conditions could distort the test results.
  3. Baseline Symptom Documentation: Before the test begins, the patient's current nasal symptoms, including congestion, rhinorrhea, sneezing, and nasal itching, are documented, preferably during asymptomatic periods.
  4. Allergen Preparation: Allergens, such as pollen, dust mites, animal dander, and molds, are prepared for the provocation. These allergens are diluted to appropriate concentrations for the test.
  5. Provocation Procedure: The allergen solution is introduced into the patient's nasal cavity, with the dosage and concentration being incrementally adjusted based on the patient's response by the overseeing physician.
  6. Symptom Observation and Documentation: Following allergen administration, the patient is monitored closely for the development of allergic symptoms. The severity and onset time of symptoms such as nasal congestion, rhinorrhea, and sneezing are recorded.
  7. Result Interpretation: The presence of allergic symptoms after provocation indicates an allergy to the introduced allergen, leading to a diagnosis of LAR.
  8. Symptom Relief: Should the patient experience significant allergic symptoms, relief may be provided through the administration of antihistamines or other appropriate medications.

     This diagnostic test is potent but requires professional medical supervision due to the inherent risk of triggering severe allergic reactions. Emergency preparedness is essential throughout the procedure to ensure patient safety.
* Nasal eosinophilic infiltration: To assess the degree of local eosinophilic infiltration in the nasal cavity, a cytological analysis of nasal secretions is performed. This involves the collection of nasal secretions from the nasal cavity using swabs. The swabs are gently inserted into the nostrils and rotated to collect the necessary sample.

Once the sample is collected, it is then subjected to cytological analysis. This analysis involves examining the nasal secretions under a microscope to identify and quantify the presence of eosinophils, which increases in number in patients with NARES.

In addition to cytological analysis, the detection of specific biomarkers such as eosinophilic cationic protein (ECP) and Charcot-Leyden crystal proteins can provide further insight into the degree of local eosinophilic infiltration and activation. ECP is a protein released by activated eosinophils and is associated with the cytotoxic activity of these cells. Charcot-Leyden crystals are hexagonal crystalloid structures that form within the secretions of eosinophils and can be identified in cytological preparations.

By combining the results of cytological analysis with the detection of these biomarkers, healthcare professionals can obtain a comprehensive assessment of the degree of local eosinophilic infiltration in the nasal cavity. This information can be useful in the diagnosis of NARES.

* Dry cold air provocation test : To assess the high reactivity of the nasal cavity to physical stimulation, particularly in the context of Idiopathic Rhinitis (IR) or other nasal hyperreactivity conditions, a local nasal cavity stimulation with dry cold air can be performed. This stimulation is designed to replicate the exposure to cold, dry air that often triggers symptoms in individuals with sensitive nasal passages. Here's a detailed description of the procedure:

  1. Preparation: Prior to the stimulation, the patient should be comfortably seated in a quiet, temperature-controlled room. It is important to ensure that the patient is not suffering from an acute upper respiratory infection or any other condition that might affect the results of the test.
  2. Equipment Setup: A device capable of delivering a controlled flow of dry cold air is used for the stimulation. The device should be able to maintain a temperature range of 5-15°C, a humidity level of 10%-15%, and a flow rate of 20-30 liters per minute, as these parameters have been determined to be provocative for individuals with hyperreactive nasal cavities.
  3. Patient Instruction: The patient is instructed to breathe normally through the nose during the procedure. They should be informed about what to expect during the stimulation and assured that the test is safe and monitored closely by the medical staff.
  4. Stimulation: The dry cold air is directed towards the patient's nostrils using a specialized nozzle.
  5. Duration: The stimulation typically lasts for a few minutes, usually between 5 and 10 minutes, depending on the patient's response. The duration can be adjusted based on the patient's tolerance and the appearance of symptoms.
  6. Symptom Monitoring: Throughout the stimulation, the patient's response is closely monitored for symptoms such as sneezing, nasal congestion, rhinorrhea (runny nose), and nasal itching. These symptoms indicate a hyperreactive response to the cold, dry air.
  7. Post-Stimulation Assessment: After the stimulation, the patient's nasal symptoms are assessed and recorded. Any relief or persistence of symptoms is noted, which can provide valuable information for the diagnosis of IR or other nasal hyperreactivity conditions.
  8. Safety Measures: It is essential to have emergency medications and equipment on hand in case the patient experiences an exaggerated reaction to the cold air stimulation.

     This procedure allows healthcare professionals to evaluate the degree of nasal hyperreactivity to physical stimuli and can help diagnose of IR.
* Peripheral blood, serum, and/or nasal mucosal epithelial cells will be collected for Proteomic detection.

ELIGIBILITY:
Inclusion Criteria:

Chinese aged between 18 and 70 years old who have resided at the survey site for more than 6 months within the 12 months preceding the survey.

Exclusion Criteria:

Exclusion criteria for questionnaire recipients: ① residents in specialized facilities (e.g., workshops, military barracks, student dormitories, nursing homes); individuals with mental or cognitive disorders (including dementia, aphasia, deafness); Exclusion criteria for nasal examination participants: ① individuals who have undergone sinus or nasal surgery, or diagnosed with sinusitis, nasal polyps, or nasal/nasopharyngeal tumors in the past year; ② patients with cystic fibrosis or primary ciliary dyskinesia; ③ residents in specialized facilities (e.g., workshops, military barracks, student dormitories, nursing homes); individuals with mental or cognitive disorders (including dementia, aphasia, deafness); (5) individuals currently under treatment for newly diagnosed tumors; ⑥ volunteers deemed unsuitable for the study by the research team.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: To estimate the incidence of chronic rhinitis in China, we calculate a sample size of roughly 9,471 patients using the formula n = (Z^2 * p * (1-p))/E^2, with Z = 1.96 for a 95% confidence level, p = 0.2 for a 20% prevalence, and E = 0.015 for a 1.5% margin of error. Our study includes recalling 3,000 patients for nasal exams, implying a need to survey 18 million subjects for a 20% incidence rate and 80% response rate. We'll use a multi-stage cluster sampling survey for 18,000 face-to-face questionnaires and distribute 132,000 electronic questionnaires to reach 30,000 chronic rhinitis patients, assuming a 20% prevalence.
Sampling Method: Probability Sample
Enrollment: 150000 (Estimated)
Dates: Start 2024-04-27 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
The prevalence chronic rhinitis within the Chinese population | 2024.04-2025.04
  The overall prevalence of chronic rhinitis across the Chinese population will be discribed. This will provide a demographic breakdown of how common chronic rhinitis is among various segments of the population.

SECONDARY OUTCOMES:
The distribution patterns of chronic rhinitis within the Chinese population | 2024.04-2025.04
  The prevalence of subtype of chronic rhinitis, including allergic rhinitis, local allergic rhinitis, Non-Allergic Rhinitis with Eosinophilia Syndrome (NARES), and Intrinsic Rhinitis (IR). The study will detail the percentage of patients suffering from each type of rhinitis within the Chinese population.
The risk factors of chronic rhinitis | 2024.04-2025.04
  The correlation of chronic rhinitis with various factors, such as environmental influences, personal occupation, genetic susceptibility, disease severity, and the methods used for diagnosis and treatment.
The clinical features and endotype of chronic rhinitis | 2024.04-2026.04
  Utilizing proteomic detection techniques, the study will analyze peripheral blood, serum, and nasal secretions to identify biological indicators associated with chronic rhinitis. These molecular markers will be correlated with the clinical classification of rhinitis, as established through epidemiological investigation and clinical assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Liu, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hosptial affiliated to Tongji Medical college of Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided
a

REFERENCES:
- [Background] Makar AB, McMartin KE, Palese M, Tephly TR. Formate assay in body fluids: application in methanol poisoning. Biochem Med. 1975 Jun;13(2):117-26. doi: 10.1016/0006-2944(75)90147-7. No abstract available.